CLINICAL TRIAL: NCT05648773
Title: COVID-19 Booster Incentives in a County-Run Health System
Brief Title: COVID-19 Booster Incentives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: J-PAL North America (Unknown)
Responsible Party: Principal Investigator, Mireille Jacobson, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UP-21-01097
Record Dates: First submitted 2022-12-08; First posted 2022-12-13 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Booster Message; Booster Message + Financial Incentive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Message Only (Experimental): Email or SMS Booster Vaccination Reminder
  Interventions: Behavioral: Messaging
- Message + Financial Incentive (Experimental): Email or SMS Booster Vaccination Reminder + Offer of a financial incentive for getting boosted in the next 2 weeks.
  Interventions: Behavioral: Messaging; Behavioral: Financial Incentive
- Control (Placebo Comparator): No message or financial incentive
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Messaging — Booster reminder message
  Arms: Message + Financial Incentive; Message Only
Behavioral: Financial Incentive — Financial Incentive for getting boosted within 2-weeks of the message
  Arms: Message + Financial Incentive
Other: Placebo — Treatment as usual; no additional message and no incentive.
  Arms: Control

SUMMARY:
The goal of this work is to understand whether small financial incentives and messaging can increase the take-up of COVID-19 boosters among patients empaneled at a county public health system. The motivation for this work is the relatively low take-up of COVID-19 boosters. In California, where our experiment is based, only 59% of the population has been boosted, with only 13% receiving the recommended bivalent booster (State of California, 2022).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 and above
2. At least one COVID-19 vaccination (primary series or monovalent booster) but no vaccination dose within the past 2-months.
3. Active phone number or email

Exclusion Criteria:

1. Opt-out of health system messaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57893 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Vaccine booster | 2 weeks
  Received a booster vaccination within 2-weeks of message.

CONTACTS AND LOCATIONS:
Locations (1):
- Contra Costa Health Plan, Martinez, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Access Criteria: Researchers can request de-identified data from Contra Costa Health Services.